CLINICAL TRIAL: NCT05298124
Title: Transcatheter Mitral Valve Repair for Inotrope Dependent Cardiogenic Shock
Acronym: MINOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210381-01T
Record Dates: First submitted 2022-02-11; First posted 2022-03-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cardiogenic Shock; Mitral Regurgitation
MeSH Terms: conditions — Shock, Cardiogenic; Mitral Valve Insufficiency | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcatheter edge-to-edge repair (Experimental): The experimental arm includes treatment in an intensive care unit with intravenous medications (e.g. vasopressors and inotropes), ventilatory support or mechanical circulatory support plus transcatheter edge-to-edge repair
  Interventions: Device: Transcatheter edge-to-edge repair
- Medical therapy (Active Comparator): Medical therapy includes treatment in an intensive care unit with intravenous medications (e.g. vasopressors and inotropes), ventilatory support or mechanical circulatory support.
  Interventions: Other: Medical therapy

INTERVENTIONS:
Device: Transcatheter edge-to-edge repair — Transcatheter edge-to-edge repair
  Other Names: MitraClip
  Arms: Transcatheter edge-to-edge repair
Other: Medical therapy — Medical treatment in an intensive care unit
  Arms: Medical therapy

SUMMARY:
Mitral regurgitation may be seen in the setting of cardiogenic shock. Transcatheter edge-to-edge repair (TEER) has been shown to improve outcomes in patients with chronic heart failure. Observational studies suggest improvements in clinical outcomes in patients with mitral regurgitation in the setting of cardiogenic shock; however, there remains a lack of randomized clinical data to support the use of TEER in cardiogenic shock.

This study will be a multicenter, open-label, randomized-controlled trial with two study arms: medical therapy and TEER. Patients admitted to the Cardiac Intensive Care Unit (CICU), Cardiac Surgery Intensive Care Unit (CSICU) or Intensive Care Units (ICU) at participating centers will be recruited.

The study aims to answer the question: "Does TEER in patients with SCAI stage C or D cardiogenic with concomitant moderate or greater mitral regurgitation improve outcomes as compared to medical therapy?"

The study hypothesis is that TEER will lead to an overall improvement in the composite outcome as compared to the medical therapy arm.

DETAILED DESCRIPTION:
Current management strategies for patients with SCAI stage C through E cardiogenic shock include management in a cardiac intensive care unit (CICU) or cardiac surgery intensive care unit (CSICU) with intravenous inotropes (i.e. medications to increase the pumping function of the heart), vasopressors (i.e. medications to increase blood pressure), ventilatory support, and/or mechanical circulatory support. Importantly, with the exception of revascularization, little data exists demonstrating the ability to alter prognosis in patients with cardiogenic shock.

Mitral regurgitation may be seen in the setting of cardiogenic shock. Transcatheter edge-to-edge repair (TEER) has been shown to improve outcomes in patients with chronic heart failure. Observational studies suggest improvements in clinical outcomes in patients with mitral regurgitation in the setting of cardiogenic shock; however, there remains a lack of randomized clinical data to support the use of TEER in cardiogenic shock.

This study will be divided into two phases, as follows:

Phase 1 (Vanguard) - The first phase of this study will be composed of a feasibility stage where a total of 10 participants from centers in Ontario, Canada will be recruited. The primary objective of this phase is to ascertain feasibility of participant recruitment and treatment. Feasibility would be considered met if 10 participants were enrolled 12 months from the date of activation of all four centers.

Phase 2 - The second phase of this study will be a continuation of Phase 1 where the remaining 134 participants, for a total of 144 participants in the overall study. For this second phase of the study, patients will be recruited from high-volume TEER centers in Canada and the United States - with participating centers performing more than 25 TEER procedures per year.

Eligible participants will be randomly assigned in a 1:1 fashion to the medical therapy arm (i.e. control arm) or the TEER arm (i.e. intervention arm) of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or substitute decision maker is able and willing to provide written informed consent
2. Age ≥ 18 years
3. SCAI stage C or D cardiogenic shock with persistent inotrope/vasopressor/non-durable mechanical support or unable to wean ventilatory support due to pulmonary edema for 24 hours prior to randomization
4. Greater than or equal to 3+ MR as determined by a study center's transesophageal echocardiogram (TEE)
5. In the opinion of the study center's heart team the participant is anatomically eligible for TMVr with the potential to achieve <3+ MR

Exclusion Criteria:

1. Unwilling or unable to obtain informed consent from the participant or substitute decision maker
2. Revascularization of coronary artery disease performed in the 48 hours prior to randomization
3. If the mechanism of MR is deemed to be degenerative, in the opinion of the heart team the participant is eligible for surgical intervention
4. Prior mitral valve leaflet surgery or implanted mitral valve prosthesis (excluding ring)
5. Echocardiographic evidence of left sided intracardiac mass or thrombus
6. Diagnosis of active infective endocarditis
7. Transesophageal echocardiogram is contraindicated
8. Mitral valve anatomy deemed contraindication to TMVr implantation that cannot be addressed procedurally as determined by the study center's heart team
9. Any aortic valve disease greater than moderate in severity
10. A known hypersensitivity or contraindication to procedure medications which cannot be adequately managed medically
11. Out of hospital cardiac arrest or in-hospital cardiac arrest without documented neurologic recovery
12. Plan for durable mechanical circulatory support implantation prior to TMVr
13. In the opinion of the treating team, there is a significant comorbidity that would limit life expectancy in hospital
14. Pregnant or planning to become pregnant in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary composite outcome | Through duration of hospitalization, generally up to 12 weeks following admission
  The primary outcome in this clinical trial will be a composite of in-hospital all-cause mortality, cardiac transplantation, implantation of durable LVAD, or discharge on palliative inotropic therapy.

SECONDARY OUTCOMES:
In hospital all-cause mortality | Through duration of hospitalization, generally up to 12 weeks following admission
  Death from any cause
In hospital implantation of durable left-ventricular assist device or cardiac transplantation | Through duration of hospitalization, generally up to 12 weeks following admission
  Implantation of durable left-ventricular assist device or cardiac transplantation
Discharge on inotropes | Through duration of hospitalization, generally up to 12 weeks following admission
  Discharge from index hospitalization on palliative inotropic therapy
Residual mitral regurgitation | Through duration of hospitalization, generally up to 12 weeks following admission
  Severity of residual mitral regurgitation as assessed by the core lab on last available in hospital echocardiogram
Technical success | Measured at exit from procedure room, generally 2 hours after implant
  All of the following must be present:
  I. Absence of procedural mortality II. Successful access, delivery, and retrieval of the device delivery system III. Successful deployment and correct positioning of the first intended device IV. Freedom from emergency surgery or reintervention related to the device or access procedure.
Device success | At time of discharge from hospitalization, generally up to 12 weeks following admission
  All of the following must be present:
  I. Absence of procedural mortality or stroke II. Proper placement and positioning of the device III. Freedom from unplanned surgical or interventional procedures related to the device or access procedure
  IV. Continued intended safety and performance of the device, including:
  A. No evidence of structural or functional failure B. No specific device-related technical failure issues and complications C. Reduction of mitral regurgitation to either optimal or acceptable levels without significant mitral stenosis, and with no greater than mild (1+) paravalvular mitral regurgitation (and without associated hemolysis)
Stroke or transient ischemic attack | Through duration of hospitalization, generally up to 12 weeks following admission
  Acute episode of a focal or global neurological deficit as determined by or in conjunction with the designated neurologist
Bleeding | Through duration of hospitalization, generally up to 12 weeks following admission
  * Any intracranial bleeding (excluding microhemorrhages <10 mm evident only on gradient-echo MRI)
  * Clinically overt signs of hemorrhage associated with a drop in hemoglobin of ≥5 g/dL or a ≥15% absolute decrease in hematocrit
  * Fatal bleeding (bleeding that directly results in death within 7 d)
Vascular access complications | Through duration of hospitalization, generally up to 12 weeks following admission
  Access site-related arterial or venous injury or injury to surrounding structures
Cardiac structural complications | Through duration of hospitalization, generally up to 12 weeks following admission
  Cardiac perforation or pseudoaneurysm

OTHER OUTCOMES:
All-cause mortality | 6 months
  Death from any cause
All-cause hospitalization | 6 months
  Hospitalization is defined as admission to an inpatient unit or ward in the hospital for ≥24 h, including an emergency department stay. Hospitalizations planned for pre-existing conditions are excluded unless there is worsening of the baseline condition.
Any re-intervention on the mitral valve | 6 months
  Requiring any transcatheter or surgical re-intervention on the mitral valve

CONTACTS AND LOCATIONS:
Locations (4):
- Mayo Clinic, Rochester, Minnesota, United States
- Canada (3):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan is to be decided upon at trial completion.